CLINICAL TRIAL: NCT04445402
Title: Retrospective and Prospective Database of COVID-19 Prevalence and Clinical Course in Pediatric and Young Adult Hematology/ Oncology/Stem Cell Therapy Patients in the New York Tri-State Area.
Brief Title: Pediatrics HOT COVID-19 Database in NY Tristate
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAT0268
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pediatric Cancer; Immune System Disorder; COVID-19; Hemoglobinopathies
Keywords: Immune System Disorder in Children; Immune System Disorder In Young Adults
MeSH Terms: conditions — Neoplasms; Immune System Diseases; COVID-19; Hemoglobinopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Optional stool specimens may be collected at three time points: 1) at diagnosis, 2) at resolution of COVID-19, 3) and at six months post-diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Heme/Non-Sickle Cell Disease: Subjects with a diagnosis of hemoglobinapathy except Sickle Cell Disease
- Heme/Sickle Cell Disease: Subjects with a diagnosis of Sickle Cell Disease
- Neuro-Oncological Disease: Oncology diagnosis with involvement of the neurological system
- Oncology/Non-Neuro-Oncological: Subjects with any oncology diagnosis except those that involve the neurological system.
- Transplant patients: Subjects who have received or are intending to have a stem cell transplant for treatment of disease.

SUMMARY:
New York City (NYC) has become the epicenter of the worldwide pandemic caused by severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). By collecting and summarizing the experience with other major health care providers in the tristate (New York (NY), New Jersey (NJ) and Connecticut (CT)) are, the investigators are uniquely positioned to inform the rest of the country about what to expect and how to manage children and young adults with hematological, oncological or stem cell transplant diagnoses during the pandemic.

DETAILED DESCRIPTION:
The subjects are all pediatric hematology, oncology or stem cell transplant (HOT) children and young adults who are tested for SARS-CoV-2. The investigators will collect data including demographics, clinical characteristics, clinical courses, outcomes from the medical record.

Other information about finances, mental health, and nutrition will be ascertained by questionnaires. The subjects will be asked to allow the researchers to abstract information from their medical record, participate in an interview or telephone call (their choice) to answer questionnaires, and to provide a stool sample at three time points.

The creation of an integrated database of COVID-19 pediatric and young adult patients will better inform the pediatric hematology, oncology, and stem cell transplant community about this disease specifically related to patients undergoing HOT therapy and provide valuable evidence to develop standardized and clinically appropriate approaches to their care.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic, Oncologic or Stem Cell Transplant Diagnosis
* Tested for COVID-19
* Age up to 21 years of age

Exclusion Criteria:

* Unwillingness to participate

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from birth to 21 years who have a hematologic, oncologic or stem cell transplant diagnosis and have been tested for COVID-19
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Number of tristate area pediatric HOT patients tested for COVID-19 that completed 1 year follow-up | One year
  To measure the success of the data registry in how many patients agreed to participate and completed the one year follow up. A confirmed case of COVID-19 is defined as a positive result on a reverse-transcriptase- polymerase-chain-reaction (RT-PCR) assay of a specimen collected on a nasopharyngeal swab, or a serum antibody test. Only laboratory-confirmed cases will be described as positive.

SECONDARY OUTCOMES:
Change in PROMIS T-score | Baseline, 3 Months, 6 Months
  To analyze effect of COVID-19 on patients and their families mental health. PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Number of collected and analyzed stool samples | Up to one year
  To examine if the pandemic has effects on the patients' nutrition and microbiome. Each patient is given an opportunity to provide stool samples in addition to survey response.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Satwani, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States